CLINICAL TRIAL: NCT05266911
Title: Home-based High Intensity Functional Strength Training (HIFST) for Older Adults: A Pilot Randomized Controlled Trial of an Exercise Program to Prevent Functional Decline After an Injury
Brief Title: Home-based HIFST for Older Adults to Prevent Functional Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Julie Richardson, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13879
Record Dates: First submitted 2022-01-28; First posted 2022-03-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Mobility Limitation; Fall Injury; Slip and Fall
Keywords: Preclinical Mobility Limitation; High-intensity Functional Strength Training; Feasibility; Physical Functioning; Cognitive Functioning; Enjoyment
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled trial and follow-up qualitative description study.
Who Masked: Outcomes Assessor
Masking Description: statistical analysis for secondary outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity strength training (HIFST) program (Experimental): Home-based high-intensity strength training program
  Interventions: Behavioral: high-intensity functional strength training
- Lower extremity stretching program (Active Comparator): Lower extremity stretching program
  Interventions: Behavioral: Lower extremity stretching

INTERVENTIONS:
Behavioral: high-intensity functional strength training — HIFST is an exercise program using an interval format: alternating periods of high intensity/'hard' exercise using everyday lower-extremity based strength-building movements (e.g., sit to stand) with periods of light/'easy' activity. High-intensity is individualized based on the use of a rating of perceived exertion (RPE) scale. The program includes a warm-up and cool-down and will be completed in participant's homes 3 days per week.
  Arms: High-intensity strength training (HIFST) program
Behavioral: Lower extremity stretching — Lower extremity stretching program to be completed by participants at home 3 days per week.
  Arms: Lower extremity stretching program

SUMMARY:
After an injury, an older adult may experience changes to how they complete their daily activities and participate in physical activity. Changes in how or how often an older adult performs an activity (such as climbing the stairs) can be warning signs of increased future difficulties. The purpose of this study is to prevent this decline by providing an exercise program for older adults experiencing these changes. This pilot study will determine if a 12-week home-based high intensity functional strength training (HIFST) program is feasible for older adults who have had an injury from a slip, trip, or fall. HIFST involves combining periods of performing 'hard' everyday movements to build strength (for example standing and sitting from a chair) with periods of rest or 'easy' activity. Feasibility will be determined based on the amount of recommended exercise sessions people complete, the ability to enroll participants and have them finish the program, as well as demonstration of safety. The study will also measure the effects on physical functioning, cognitive functioning, and enjoyment. Interviews with participants in the HIFST program will be conducted after the 12-weeks to gather information on their experience, opinions, likes/dislikes, and suggestions. All this information will be used to guide a future larger study to determine effectiveness.

DETAILED DESCRIPTION:
An injury from a slip, trip or fall in an older adult may instigate the onset of preclinical mobility limitation (PCML) which is a period of time in which modifications in task performance are indicative of an early stage of functional decline. Effective and enjoyable exercise interventions, which may be offered by home-based high-intensity functional strength training (HIFST), are needed during this period. More research is needed on the feasibility of conducting a home-based HIFST in a this group as well it's effects on physical functioning, cognitive functioning and enjoyment. This information, in conjunction with follow-up interviews to asses acceptability, will be used to inform plans of a future fully-powered trial to assess effectiveness.

The primary objective of this trial is to determine the feasibility of 12 weeks of home-based HIFST for community-dwelling older adults who are post-injury as determined by adherence, recruitment, retention, and safety criteria. The secondary objectives are to determine preliminary evidence of effects on physical functioning, cognitive functioning (specifically executive functions and processing speed) and physical activity enjoyment. The investigators will also report any intervention-related adverse events (harms, such as muscle strains, sprains, etc.). The follow-up qualitative study will assess acceptability of the intervention including barriers/facilitators to participation and recommendations for changes.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking, community-dwelling older adults ≥ 55 years, who
2. sustained an injury from a slip, trip or fall in the last year (assessed by self-report) and
3. as a result report decreased and/or modified daily task performance (assessed using PCML questionnaire based on Mänty) and Participants must have
4. no contraindications to exercise based on the American College for Sports Medicine recommendations and 5) complete the Canadian Society for Exercise Physiology (CSEP) 'Get Active' questionnaire and obtain clearance from a health care professional if deemed necessary based on screening.

6) Participants will be required to have access to email and a laptop/tablet with webcam capable of running the web-based videoconferencing platform Zoom well as 7) the ability to provide informed consent.

Exclusion Criteria:

1) a score of < 11 on the Mini Montreal Cognitive Assessment (Mini MoCa).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Feasibility: Adherence | over 12 weeks (intervention duration)
  Percentage of exercise sessions completed (criteria: at least 70 precent)
Feasibility: Recruitment | 4-6 month recruitment period
  Percentage of eligible participants recruited (criteria: at least 65 precent)
Feasibility: Retention | over 12 weeks
  Percentage of participants completing baseline and follow-up assessments (criteria: at least 80 percent)
Feasibility: Safety (number/presence of intervention-related serious adverse events) | over 12 weeks (intervention period)
  Adverse events related to intervention (criteria: no serious events)

SECONDARY OUTCOMES:
Physical Functioning: 4 meter walk test ( | pre and post intervention (12 weeks)
  usual gait speed over 4 meters
Physical Functioning: dual-task cognitive Timed Up and Go (TUG-COG) | pre and post intervention (12 weeks)
  time to rise from a standard chair, walk 3 meters, turn around, walk back to the chair and sit down while counting backwards by three
Physical Functioning: Two minute step test (TMST) | pre and post intervention (12 weeks)
  number of steps in two minutes
Physical Functioning: 30-second chair stand test (30CST) | pre and post intervention (12 weeks)
  number of full stands from a chair in 30 seconds
Physical Functioning: Preclinical Mobility Limitation (PCML) scale | pre and post intervention (12 weeks)
  classified as no mobility limitation, preclinical mobility limitation, minor manifest limitation or major manifest limitation for 3 tasks (walking 0.5km, walking 2 km, and climbing one flight of stairs)
Cognitive Functioning: California Older Adult Stroop Test (COAST) | pre and post intervention (12 weeks)
  measures executive functioning by assessing the ability to inhibit an automatic response
Cognitive Functioning: Digit Symbol Substitution Test (DSST) | pre and post intervention (12 weeks)
  assesses various aspects of cognition, including processing speed and several aspects of executive functioning (planning, attention, and working memory)
Cognitive Functioning: Oral Trail Making Test (OTMT) | pre and post intervention (12 weeks)
  involves task-shifting (mental flexibility), attention, working memory and processing speed
Enjoyment: Physical Activity Enjoyment Scale (PACES) | week 1,2,4,6,8,10,12
  Scale 8-56 (higher score is greater enjoyment)
Affective response to exercise: Feelings Scale (FS) | week 1,2,4,6,8,10,12
  Scale +5 to -5 (+5 very good, -5 very bad)
Harms | over 12 week intervention period
  any intervention-related adverse events (e.g., muscle soreness, muscle strains, etc.,) reported by participants

OTHER OUTCOMES:
Process Outcome: Self Efficacy for Exercise Scale (SEE) | pre and post intervention (12 weeks)
  Scale 0-90 (higher scores is greater self-efficacy)
Process Outcome: Activities Balance Confidence (ABC) Scale | pre and post intervention (12 weeks)
  0-100 percent, higher scores equals greater confidence

CONTACTS AND LOCATIONS:
Overall Officials: Julie Richardson, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No